CLINICAL TRIAL: NCT02796352
Title: A Phase II Study of High Dose Bolus IL2 in Patients With Inoperable Stage III or Stage IV Melanoma Who Have Failed Prior Anti-PD1 Immunotherapy: Efficacy and Biomarker Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Ahmad Tarhini (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-114
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High dose bolus interleukin-2 (HD IL2) (Experimental)
  Interventions: Drug: High dose bolus interleukin-2 (HD IL2)

INTERVENTIONS:
Drug: High dose bolus interleukin-2 (HD IL2) — Each course consists of 2 cycles of HD IL2 as follows: high-dose IL2 at 600,000 IU/kg is given intravenously (IV) every 8 hours for up to 14 doses (one cycle), followed by a rest period of 1-2 weeks and readmission for a second HD IL2 cycle for up to 14 doses (second cycle).
  The planned treatment consists of 3 courses (6 cycles) of HD IL-2.

SUMMARY:
This study is for patients with advanced stage III or stage IV melanoma not adequately treated by surgery who have progressed after treatment with nivolumab or pembrolizumab. The purpose of this study is to see if giving high dose interleukin-2 (IL-2) after progression on nivolumab or pembrolizumab is effective in treating metastatic melanoma. This study is also being done to look at the severity of side effects of IL-2 in patients.

IL-2 is approved by the U.S. Food and Drug Administration (FDA) for the treatment of advanced melanoma.

DETAILED DESCRIPTION:
This is a phase II study of high dose bolus interleukin-2 (HD IL2) in patients with advanced inoperable stage III or stage IV melanoma who have prior anti-PD1 immunotherapy.

Each course consists of 2 cycles of HD IL2 as follows: high-dose IL2 at 600,000 IU/kg is given intravenously (IV) every 8 hours for up to 14 doses (one cycle), followed by a rest period of 1-2 weeks and readmission for a second HD IL2 cycle for up to 14 doses (second cycle).

The planned treatment consists of 3 courses (6 cycles) of HD IL-2. Response assessment will occur at the end of each course of therapy and patients without evidence of disease progression (Response Evaluation Criteria in Solid Tumors, RECIST, version 1.1) or limiting toxicities will be offered additional courses of treatment of HD IL2 for a maximum of 3 courses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic melanoma. This includes American Joint Committee on Cancer (AJCC) stage IV or advanced/inoperable stage III. This also includes patients with a history of lower stage melanoma and subsequent recurrent metastatic disease that is either locally/regionally advanced/inoperable disease or distant metastases.
* Patients must have measurable disease, according to RECIST version 1.1
* Patients must be free of active brain metastasis by contrast-enhanced CT/MRI scans within 4 weeks prior to enrollment. If known to have prior brain metastases, these must have been adequately managed with standard of care radiation therapy, stereotactic radiosurgery or surgery prior to registration on the study.
* A patient must have previously received anti-PD1 immunotherapy (nivolumab or pembrolizumab) and later experienced disease progression, within 3 months of registration on this study.
* Patients must not have received systemic therapy or radiotherapy within the preceding 3 weeks. Patients must have recovered from adverse events from previous therapy by the time registration.
* Patients must be at least 4 weeks from major surgery and have fully recovered from any effects of surgery, and be free of significant detectable infection prior to registration.
* For patients who have received prior anti-CTLA4 monoclonal antibody therapy (ipilimumab or tremelimumab), there is a risk of bowel perforation with IL-2 therapy. Therefore, for these patients if they have a history of colitis or diarrhea during anti-CTLA4 monoclonal antibody therapy, it is recommended that they have a formal evaluation by a gastroenterologist and a colonoscopy/endoscopy should be considered to demonstrate the absence of active bowel inflammation before initiating IL-2 therapy on this protocol.
* Life expectancy of greater than 3 months in the opinion of the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >/=70%)
* Patients must have normal organ and marrow function as defined in the clinical trial protocol.
* Patients on full-dose anticoagulants (e.g., warfarin) with prothrombin time (PT)/ international normalized ratio (INR) >1.5 are eligible provided that both of the following criteria are met: (a) The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin. (b) The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices).
* Pulmonary: forced expiratory volume at one second (FEV1) > 2.0 liters or > 75% of predicted for height and age. Pulmonary function tests (PFTs) are required for patients over 50 years old or with significant pulmonary or smoking history.
* Cardiac: No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than 6 months prior to entry, serious cardiac arrhythmias, or unstable angina. Patients who are over 40 years old or have had previous myocardial infarction greater than 6 months prior to study entry or have significant cardiac family history (CAD or serious arrhythmias) will be required to have a negative or low probability cardiac stress test (for example, thallium stress test, stress multigated acquisition (MUGA), stress echo or exercise stress test) for cardiac ischemia within 8 weeks prior to registration.
* Central Nervous System (CNS): No history of cerebrovascular accident or transient ischemic attacks within the past 6 months from registration.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after completion of study therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Women should not be lactating and, if of childbearing age, should have a negative pregnancy test (b-HCG test; serum or urine, minimum sensitivity 25 IU/L or equivalent units of b-HCG) within two week of registration in the study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had systemic therapy for melanoma or radiotherapy within 3 weeks prior to registering on the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier. Patients with a history of endocrinopathies (e.g. hypothyroidism, adrenal insufficiency, hypopituitarism) are eligible if they are stable on hormone replacement therapy.
* Patients may not be receiving any other investigational agents.
* Patients with active brain metastases should be excluded from this clinical trial except as noted above.
* Patients with clinically significant cardiovascular or cerebrovascular disease:

  1. history of cerebrovascular accident or transient ischemic attack within past 6 months from registration.
  2. myocardial infarction, coronary artery bypass grafting (CABG) or unstable angina within the past 6 Months from registration.
  3. New York Heart Association grade III or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris within past 6 months from registration.
  4. clinically significant peripheral vascular disease within past 6 months from registration.
* PT INR >1.5 unless the patient is on full-dose warfarin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have other current malignancies are not eligible. Patients with other malignancies are eligible if they have been continuously disease free for > 2 years prior to the time of registration. Patients with prior history at any time of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or melanoma in situ are eligible. Patients with prior history of basal or squamous skin cancer are eligible. Patients who have had multiple primary melanomas are eligible.
* Patients must not have autoimmune disorders or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids or steroid inhalers. If a patient had been taking steroids, at least 2 weeks must have passed since the last dose. Patients stable on physiologic replacement doses of steroids or other forms of hormone replacement therapy are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 63 [63 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of complete responses (CR) plus partial responses (PR), based upon Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Time Frame: Up to 15 months for accrual, plus 6 months of intervention for last subject enrolled (21 months)
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of months of survival without disease progression from start of protocol therapy until objective tumor progression or death, per RECIST v1.1
Time Frame: Up to 15 months for accrual, plus 6 months of intervention for last subject enrolled, plus 5 years of follow-up (6 years, 9 months)
Measure: Number; unit: months
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Number analyzed (Participants) | 1
months | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Number of months from start of protocol therapy until death from any cause.
Time Frame: as for outcome 2
Measure: Number; unit: months
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Number analyzed (Participants) | 1
months | 4

4. Secondary Outcome: HD IL2 Levels
Description: Levels of HD IL2 biomarker in the blood of patients that received at least course 1 of therapy, and have had their disease re-evaluated will be considered evaluable for response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) version 1.1
Time Frame: Up to 21 months
Population: No data displayed because data were not collected for this Outcome Measure, thus zero total participants analyzed.
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From study entry until end of treatment (4 months)
Arm/Group | High Dose Bolus Interleukin-2 (HD IL2)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Bolus Interleukin-2 (HD IL2) (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT02796352/Prot_SAP_000.pdf